CLINICAL TRIAL: NCT01440777
Title: Effectiveness and Adherence to an Online Sleep Program - A Pilot Study
Brief Title: Effectiveness and Adherence to an Online Sleep Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Linda Libertini, Research Coordinator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB# 11-860
Record Dates: First submitted 2011-09-23; First posted 2011-09-27 (Estimated); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Insomnia
Keywords: Insomnia; Sleep; Stress; Online program; Web-based program; Cognitive Behavioral Therapy for Insomnia (CBT-i)
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Go! to Sleep (Active Comparator): Participants access and utilize the 6-week online program that provides a set of various psycho-educational materials and behavioral techniques to treat insomnia.
  Interventions: Behavioral: Go! to Sleep
- Control Group (No Intervention): No intervention provided. These participants will receive the Go! to Sleep program after the research trial has been completed (10 weeks after registration).

INTERVENTIONS:
Behavioral: Go! to Sleep — The online program provides various tools for the delivery of the intervention including:
  * Daily articles
  * Daily activities to help get the sleep you need
  * Daily sleep improvement recommendations
  * Audio recorded relaxation exercises
  * Daily e-mails from your program coach
  * Personal progress charts
  * An online sleep log and daily sleep score
  Arms: Go! to Sleep

SUMMARY:
This research will examine the effectiveness of a 6-week online sleep program (Go! To Sleep) which provides a set of various psycho-educational materials and behavioral techniques to reduce insomnia symptoms, improve sleep, and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years old.
* Currently living in the continental United States and Canada.
* Symptoms of insomnia based on the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) definition of insomnia disorder:

  * Self-reported sleep difficulties (including sleep-onset latency, waking after sleep onset, early waking of more than 30 min duration) 3 or more times a week in the past 3 months.
  * Self-reported insomnia problem for more than 3 months.
  * Self-reported significant daytime impairment due to sleep difficulties.
* Willingness to log onto the internet on a regular basis for the duration of the study (3-7 months).
* Willingness and able to complete almost daily a sleep log to track sleep pattern for up to 2 months at a time (approximately 2-3 min daily).
* Willingness to be in the Wait-list control group and not have access to the program for 3 months.

Exclusion Criteria:

* Pregnant or planning to be pregnant in the next 6 months.
* Lack of internet access and/or Mac computer at place of residence.
* Currently participating or have participated in group or individual therapy for insomnia in the prior month.
* Patient Health Questionnaire (PHQ9) depression score >14.
* Recent treatment (less than 3 months) or medication for depression or anxiety.
* Change in treatment or medication for depression or anxiety in the past month or planned change in the next 3 months.
* Current treatment (therapy, prescription) for any other psychological or emotional conditions (including but not limited to: mania, manic-depression, psychosis, schizophrenia, adjustment disorder).
* Diagnosed and currently suffering from a sleep disorder (including, but not limited to sleep apnea, restless leg syndrome, sleep walking, narcolepsy) which is untreated or has been treated for less than a month.
* Suffer from physical symptoms or medical conditions that may affect sleep (including but not limited to: pain, arthritis, tinnitus, diabetes, night time cough, shortness of breath, hot flashes, frequent urination, heartburn).
* Steroid an stimulant use (including but not limited to prednisone, methylprednisolone or Solumedrol (for inflammatory disorders), methylphenidate, or Ritalin (for Attention-Deficit Hyperactivity disorder), Provigil (for narcolepsy), Wellbutrin or Zyban (for tobacco cessation), cocaine or methylenedioxymethamphetamine (MDMA) (a.k.a. Ecstasy)).
* Irregular workshift.
* Having young children who may affect sleep pattern.
* Taking over-the-counter or prescribed sleep medication 3 or more times a week.
* Alcoholism.
* Inability to access the internet on a consistent regular basis for the duration of the study (3-7 months).
* Inability to complete daily sleep log to track sleep patterns for up to 2 months at a time.
* Unwillingness to be assigned to the wait-list control group for 3 months prior to gaining access to the program.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2011-10; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Insomnia severity | 5 months
  To assess the effectiveness of the online Go! to Sleep program in improving sleep by measuring insomnia severity using the Insomnia Severity Index (ISI).

SECONDARY OUTCOMES:
Insomnia symptoms | 5 months
  To determine if the program helps improve insomnia symptoms as measured by the Pittsburgh Insomnia Rating Scale (PIRS)
Sleep pattern | 5 months
  To determine if the program helps improve sleep-onset latency (SOL), total sleep time (TST), waking after sleep onset (WASO) (within Go To Sleep! group analysis only)
Daytime Dysfunction | 5 months
  To determine if the program improves daytime dysfunction (Pittsburgh Sleep Quality Index subscale)
Stress | 5 months
  To assess whether the program reduces stress as measured by the Perceived Stress Scale (PSS10)
Program adherence | 5 months
  To assess program adherence and its relation to program effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Adam Bernstein, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States